CLINICAL TRIAL: NCT07166692
Title: Evaluation of a Retrieval Augmented Large Language Model as a Diagnostic Copilot in Rheumatology
Acronym: ALLIANCE
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Philipps University Marburg (Other)
Collaborators: University Medical Center Hamburg-Eppendorf (UKE) (Unknown); Oslo University Hospital (Other); Diakonhjemmet Hospital (Other); University Hospital Erlangen (Other); Charite University, Berlin, Germany (Other); Rheumazentrum Ruhrgebiet (Other); University of Lausanne Hospitals (Other); Klinikum Fulda (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: 24-221-1
Record Dates: First submitted 2025-08-25; First posted 2025-09-10 (Actual); Last update posted 2025-09-10 (Actual); Status verified 2025-09

CONDITIONS: Diagnosis
Keywords: Clinical reasoning; Large language models; Computer-assissted diagnosis; Rheumatology
MeSH Terms: conditions — Disease

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: The evaluation of responses will be performed by assessors blinded to participant identity and treatment assignment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Prof. Valmed (Experimental): Group will be given access to Prof. Valmed.
  Interventions: Other: Prof. Valmed
- Control group (No Intervention): Group will not be given access to Prof. Valmed but will be encouraged to use any resources they wish besides large language models (UpToDate, etc).

INTERVENTIONS:
Other: Prof. Valmed — Prof Valmed. decision support system.
  Arms: Prof. Valmed

SUMMARY:
This trial evaluates whether providing physicians with access to Prof. Valmed, a clinical decision support medical product, improves identification of rheumatic diseases and formulation of differential diagnoses compared with conventional decision support.

DETAILED DESCRIPTION:
Advanced AI, particularly large language models, shows promise for enhancing clinical reasoning, yet most systems such as ChatGPT are not certified as medical products. Prof. Valmed is a clinical decision support medical product designed to assist physicians in diagnostic decision making. Given frequent referral problems and diagnostic delays in rheumatology, evaluating such support is highly relevant for clinical workflows.

This randomized controlled trial will test whether access to Prof. Valmed improves physicians' diagnostic performance in cases of suspected rheumatic disease compared with conventional decision support. Participants will be randomized to either use Prof. Valmed or rely on conventional tools while working through standardized clinical cases. For each case, participants will submit up to three differential diagnoses and a confidence rating. Independent reviewers, blinded to group allocation, will adjudicate accuracy. Findings will clarify the benefits and limitations of integrating Prof. Valmed into routine practice.

ELIGIBILITY:
Inclusion Criteria:

* Participants must be licensed physicians.
* Training in rheumatology, internal medicine, emergency medicine, family medicine, dermatology or orthopedics.

Exclusion Criteria:

* Not currently practicing clinically.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 82 (Estimated)
Dates: Start 2025-10-02 (Estimated); Primary Completion 2026-02-02 (Estimated); Study Completion 2026-02-02 (Estimated)

PRIMARY OUTCOMES:
Diagnostic accuracy of top diagnosis | directly (within 10 minutes) after Intervention
  Participants in each group will make at least one disease suggestion (top diagnosis) and up to a total of a maximum of 3 suggestions. Percentage of exact matches of the top suggestion with the actual diagnosis will be analyzed

SECONDARY OUTCOMES:
Diagnostic accuracy of top 3 suggestions | directly (within 10 minutes) after Intervention
  Participants in each group will make at least one disease suggestion (top diagnosis) and up to a total of a maximum of 3 suggestions. Percentage of exact matches with the actual diagnosis included in the top 3 suggestions will be analyzed
Diagnostic confidence | directly (within 10 minutes) after Intervention
  For each case participants will be asked for their diagnostic confidence (VAS 0-10). The mean score will be compared between groups.
Time spent for diagnosis | directly (within 10 minutes) after Intervention
  We will compare how much time (in seconds) participants spend per case between the two study arms.
Perceived Information Timeliness | directly (within 10 minutes) after Intervention
  Perceived ability to receive the information needed without delay (Likert scale from 1 to 5)
Perceived diagnostic support quality | directly (within 10 minutes) after Intervention
  Perceived quality of the diagnostic support (Likert scale from 1 to 5)
Diagnostic reasoning | during evaluation
  For each case, participants will receive 1 point for each plausible diagnosis and 2 points for a completely correct response. The total scores will be compared between the randomized groups.

CONTACTS AND LOCATIONS:
Overall Officials: Johannes Knitza, MD PhD, Principal Investigator — University Marburg
Locations (1):
- Institute for Digital Medicine, University Hospital of Giessen and Marburg, Philipps University Marburg, Marburg, Germany

IPD SHARING:
Plan to Share IPD: No